CLINICAL TRIAL: NCT06116578
Title: A Window of Opportunity (WoO) Study Evaluating Pembrolizumab With or Without Olaparib in Tertiary Lymphoid Structures (TLS)-Positive Selected Resectable Soft Tissue Sarcoma (STS) Followed by Adjuvant Pembrolizumab
Brief Title: Study Evaluating Pembrolizumab +/- Olaparib in TLS Positive Selected Resectable STS Followed by Adjuvant Pembrolizumab
Acronym: NeoSarc
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Abandon of the study by the partenair (MSD)
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-513469-38-00; 2023/3610 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2023-10-18; First posted 2023-11-03 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: sarcoma; TLS; Liposarcoma; immunotherapy; PARP
MeSH Terms: conditions — Neoplasms; Sarcoma; Liposarcoma | interventions — pembrolizumab; olaparib; Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Pembrolizumab before surgery (Active Comparator): Before surgery: Pembrolizumab 200 mg two intravenous (IV) infusions q3w (2 injections: at C1D1 and C1D21)
  Interventions: Drug: Pembrolizumab; Drug: Pembrolizumab adjuvant
- B: Pembrolizumab + olaparib before surgery (Active Comparator): Before surgery: Pembrolizumab 200 mg two IV infusions q3w (2 injections: at C1D1 and C1D21) + concomitant full dose olaparib (300 mg per os b.i.d) during four weeks
  Interventions: Drug: Pembrolizumab and Olaparib; Drug: Pembrolizumab adjuvant

INTERVENTIONS:
Drug: Pembrolizumab — cf Arm A
  Other Names: WOO (Windows of opportunity)
  Arms: A: Pembrolizumab before surgery
Drug: Pembrolizumab and Olaparib — cf Arm B
  Other Names: WOO (Windows of opportunity)
  Arms: B: Pembrolizumab + olaparib before surgery
Drug: Pembrolizumab adjuvant — After surgery (adjuvant phase), all patients (Arm A and B) will receive pembrolizumab 200 mg two intravenous (IV) infusions q3w for one-year
  Other Names: Adjuvant

SUMMARY:
Soft tissue sarcomas represent a subtype of cancer that is both rare and very heterogeneous. When they are organized, their current treatment is essentially based on tumor resection surgery, +/- associated with treatment by chemotherapy and/or radiotherapy. The aim of this treatment is to reduce the risk of local recurrence (appearance of a tumor in the same region where it was first detected) and/or distant (appearance of a tumor in other regions, organs where it was first detected).

Currently, no immunotherapy treatment has been approved for the treatment of patients with sarcoma.

This research is based on the hypothesis that soft tissue sarcomas in which "tertiary lymphoid structures" or "TLS" are found, recognizable by a cluster of specific immune cells within the tumor, would be likely to respond better to the immunotherapy. Furthermore, the combination of immunotherapy and certain drugs targeting DNA repair has demonstrated some effectiveness in other types of cancers.

Trial population :Adult patients with suspected / diagnosed soft tissue sarcoma of the extremities or trunk (Cohort 1: Undifferentiated pleomorphic sarcoma / Cohort 2: Dedifferentiated liposarcoma)

The research will therefore focus on two experimental drugs :

* Pembrolizumab (immunotherapy) and
* Olaparib (DNA repair inhibitor).

This research will make it possible to evaluate the effectiveness and safety of use of the two drugs.

DETAILED DESCRIPTION:
This study will allow:

* To evaluate the ability of pembrolizumab (with or without olaparib) before surgery to trigger an immune reaction in order to kill tumor cells.
* To evaluate the feasibility of therapy with pembrolizumab for 1 year (with or without radiotherapy) after surgery.

The research is divided into two groups of patients, called "cohorts" depending on the type of soft tissue sarcoma you have:

* Cohort 1: Undifferentiated pleomorphic sarcoma
* Cohort 2: Dedifferentiated liposarcoma

Before surgery, a group of patients will receive pembrolizumab combined with olaparib, a second group will receive only pembrolizumab. All patients will receive pembrolizumab after surgery (for up to 1 year).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years at time of informed consent signature
* Histologically confirmed diagnosis of high grade (FNCLCC grade 2 or 3) extremity, retroperitoneal, or trunk wall STS of selected histotypes as defined below. Diagnosis must be stated in a pathology report and confirmed by the physician investigator:

Cohort 1: Undifferentiated Pleomorphic Sarcoma (UPS) Cohort 2: Dedifferentiated Liposarcoma (ddLPS)

* R0 resectability at time of enrollment according to expert STS surgeon
* Absence of distant metastasis on screening CT-scan (or equivalent appropriate imaging technique)
* Patients with local relapse after an initial surgical resection can be enrolled if no perioperative chemotherapy or radiation has been previously performed Identification of Tertiary Lymphoid Structures (TLSs) on tumor archival FFPE sample, as assessed by a registered STS expert senior pathologist
* Primary tumor site measurable according to RECIST v1.1 as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and suitable for repeated assessment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no deterioration from registration date
* Adequate hematologic and organ function, defined by the following laboratory results obtained within 3 days prior to the first study treatment (Cycle 0 Day 1): Absolute neutrophil count (ANC) ≥ 1500 cells/μL, Platelet count ≥ 100.000/μL, Hemoglobin ≥ 10 g/dL, Total bilirubin ≤ 1.5 ULN (subjects with documented/suspected Gilbert's disease may be enrolled with bilirubin ≤ 3 × ULN), Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x upper normal limit (ULN), Albumin ≥ 28g/L, Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 30 mL/min (according to Cockcroft and Gault formula), International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN. This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular weight heparin or warfarin) should be on stable dose.
* Hepatitis B and C, and HIV screening tests are not required unless

  * Known history of HBV, HCV or HIV infection
  * As mandated by local health authority
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP) OR
  2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for 120 to 180 days (corresponding to time needed to eliminate any study treatment(s) plus the duration of a menstruation cycle: 120 days for pembrolizumab and/or 180 days for olaparib) after the last dose of study treatment.

Male participants:

A male participant must agree to use a contraception - Contraceptive Guidance and Pregnancy Testing of this protocol during the treatment period and for at least 180 to 240 days, corresponding to time needed to eliminate any study treatment(s) plus the duration of a spermatogenesis cycle: 180 for pembrolizumab and/or 240 days for olaparib) after the last dose of study treatment and refrain from donating sperm during this period.

* Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
* Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed.
* Patient should be able and willing to comply with baseline mandatory biopsy, as well as study visits and procedures as per protocol.
* Patients must be affiliated to a social security system or beneficiary of an equivalent system.

Exclusion Criteria:

* Has a visceral STS primary site.
* Has a non-resectable or marginally resectable locally advanced STS, as assessed by expert STS surgeon.
* Has evidence of metastatic disease on CT-scan (or equivalent imaging technique).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to randomization.
* Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids.
* Has had previous exposure to anti-PD-1, anti-PD-L1, anti-PD-L2 agent or with an agent directed to another stimulatory or co inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
* Had had previous exposure to olaparib or any other PARP inhibitor.
* Has received a live vaccine or live-attenuated vaccine received within 4 weeks prior to Cycle 0 Day 1 or anticipation that such a live attenuated vaccine will be required during the study. Administration of killed vaccines is allowed.
* Has received treatment with systemic immunostimulatory agents (e.g., IFN and IL-2) within 4 weeks prior to Cycle 0 Day 1.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has had an administration of colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior to Cycle 0 Day 1.
* A WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization (see Appendix 3 - Contraceptive Guidance and Pregnancy Testing). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has a history of severe allergic, anaphylactic, or other hypersensitivity reactions to the components of excipients in pembrolizumab and/or olaparib.
* Has any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) or immunodeficiency
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (e.g.., thyroxine, insulin, or physiologic corticosteroid)
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has a history of allogeneic tissue/organ or hematopoietic stem cell transplantation.
* Has a history of another primary malignancy within 2 years prior to Cycle 0 Day 1
* Has a serious, uncontrolled medical disorder
* Is unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption (e.g., gastrectomy, partial bowel obstruction, and malabsorption).
* Has concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA), Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection, HIV (defined as detectable viral load)
* Has any active infection requiring systemic therapy.
* Major surgical procedure within 20 days prior ty Cycle 0 Day 1 or anticipation of need for a major surgical procedure during the course of the study.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Participant is currently receiving either strong (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil) inhibitors of cytochrome P450 (CYP)3A4 that cannot be discontinued for the duration of the study. The required washout period prior to starting olaparib is 2 weeks. The medication can be restarted as soon as olaparib has been halted.
* Participant is currently receiving either strong (phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate (e.g., bosentan, efavirenz, modafinil) inducers of CYP3A4 that cannot be discontinued for the duration of the study. The required washout period prior to starting olaparib is 5 weeks for phenobarbital and 3 weeks for other agents. The medication can be restarted as soon as olaparib has been halted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Rate of CD8+ T-cell tumor infiltration density at surgery compare to baseline | 1 year after the end of inclusions
  50% increase in CD8+ T-cell tumor infiltration density between baseline biopsy and resection surgery specimen as defined by expert pathologist who will be blinded for treatment arm and patient outcome

SECONDARY OUTCOMES:
Proportion of patients with 70% pathological response | Through study completion, an average of 1 year
  Proportion of patients with 70% pathological response on the resection surgery specimen as assessed by expert pathologist after WoO treatment
Surgery evaluation: Quality of resection as defined by Hemanek and Wittekind (R0 the best / R1 / R2 the worst) | Through study completion, an average of 1 year
  Quality of resection is defined at time of resection surgery as follows, as initially defined by Hemanek and Wittekind according to both clinical and pathological findings: R0 corresponds to resection for cure or complete remission. R1 to microscopic residual tumor, R2 to macroscopic residual tumor.
Surgery evaluation : amputation rate | Through study completion, an average of 1 year
Surgery evaluation : Incidence of acute wound complications up to 120 days after surgery | 120 days after surgery
Objective Response Rate (ORR) | At 4 weeks of WoO treatment
  Objective Response Rate (ORR) at 4 weeks of WoO treatment defined as the rate of patients with Complete Response (CR) or Partial Response (PR) according to RECIST v1.1
Time To Relapse (TTR) | From date of randomization until the date of first documented Progression or date of death from any cause, whichever came first, assessed up to 75 months
Local Recurrence Rate (LRR) | 2-year post-surgery
  Local Recurrence Rate (LRR) at 2-year post-surgery
Disease Free Survival (DFS) at 2-year post-surgery | 2-year post-surgery
  Disease Free Survival (DFS) at 2-year post-surgery
Overall Survival (OS) | Through study completion, an average of 1 year
Disease Control Rate (DCR) | At 4 weeks of WoO treatment
  Disease Control Rate (DCR) at 4 weeks of WoO according to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No